CLINICAL TRIAL: NCT00059930
Title: A Phase I Study Of Hepatic Arterial Infusion With Floxuridine And Dexamethasone In Combination With Intravenous Oxaliplatin Plus 5-Fluorouracil And Leucovorin As Adjuvant Treatment After Resection Of Hepatic Metastases From Colorectal Cancer
Brief Title: Adjuvant Hepatic Arterial Infusion and Combination Chemotherapy in Treating Patients With Resectable Hepatic Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-005; MSKCC-03005
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Dexamethasone; Floxuridine; Fluorouracil; Leucovorin; Oxaliplatin; Chemotherapy, Adjuvant

ARMS (1):
- Adjuvant Hepatic Arterial Infusion & Combination Chemotherapy (Experimental): This is a Phase I study with the primary objective of defining the maximum tolerated dose of hepatic arterial floxuridine (FUDR) and dexamethasone (Dex) given via an implanted pump in combination with intravenous oxaliplatin plus systemic fluorouracil (5FU)/leucovorin (LV) in the adjuvant setting after resection of hepatic metastases from colorectal cancer. A total of eleven dose levels will be considered.
  Interventions: Drug: FOLFOX regimen; Drug: dexamethasone; Drug: floxuridine; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: adjuvant therapy; Procedure: conventional surgery

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: dexamethasone
Drug: floxuridine
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: conventional surgery

SUMMARY:
The purpose of this study is to find the highest dose that can be given safely to people who have had liver disease resected. This is a Phase I study. The goal of a phase I study is to find a safe dose range based on side effects. The drugs that will be given by vein are OXALIPLATIN ("Oxali") plus 5-FLUOROURACIL and LEUCOVORIN ("5FU" and "LV"). This is systemic chemotherapy, since it goes to the whole body. The drugs that will be placed in the pump are FLOXURIDINE (FUDR) and DEXAMETHASONE. (The dexamethasone is not an anti-tumor drug; it helps protect healthy liver tissue from possible side effects of the FUDR.) This is the regional chemotherapy, since it goes only to the liver. The researchers have studied these drugs and know the best doses of each when they are used in patients who have not had liver resections. We do not yet know how the drugs work with each other in patients with a liver resection. This study will tell us the best doses of each drug when they are given over the same period of time.

ELIGIBILITY:
Subject Inclusion Criteria:

* History of histologically confirmed colorectal adenocarcinoma metastatic to the liver with no clinical or radiographic evidence of extrahepatic disease. Confirmation of diagnosis must be performed at MSKCC.
* Potentially completely resectable hepatic metastases without current evidence of other metastatic disease.
* Abdominal and pelvic CT scans and chest CT or x-ray within 6 weeks prior to registration. (MRI of abdomen may be substituted for CT of abdomen.)
* Lab values within 14 days prior to registration:
* WBC ≥ 3.0 K/ul
* ANC >1.5 K/ul
* Platelets ≥ 100 K/ul
* Total bilirubin ≤ 1.5 mg/dl.
* Prior chemotherapy is acceptable if last dose given ≥ 3 weeks prior to registration to this study.
* KPS ≥ 60%
* Signed informed consent.

Subject Exclusion Criteria:

* Prior radiation to the liver. (Prior radiation therapy to the pelvis is acceptable if completed at least 4 weeks prior to registration.)
* Active infection, ascites, hepatic encephalopathy
* Prior oxaliplatin or cisplatin or HAI FUDR
* Female patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 2 years
Correlate thymidylate synthase, dihydropyrimidine dehydrogenase, and ERCC-1 with survival and recurrence as measured by normal and tumor liver tissue | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E. Kemeny, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/